CLINICAL TRIAL: NCT00602563
Title: Attention Training for Generalized Anxiety Disorder (Attention Training and Relaxation for GAD: Testing the Efficacy of Home-Delivery)
Brief Title: Attention Training for Generalized Anxiety Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Nader Amir, Professor, San Diego State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5R01MH087623-04 (NIH); 5R01MH087623-04 (NIH); R01MH087623 (NIH)
Record Dates: First submitted 2008-01-15; First posted 2008-01-28 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Generalized Anxiety Disorder
Keywords: Generalized Anxiety Disorder; Information Processing
MeSH Terms: conditions — Generalized Anxiety Disorder | interventions — Adenosine Monophosphate; Clinical Trials Data Monitoring Committees

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 Attention Modification Program (AMP) (Experimental): The AMP is a computer-delivered attention modification
  Interventions: Behavioral: AMP
- Applied Relaxation (AR) (Active Comparator): Applied Relaxation (AR) is a behavioral, skills-based intervention where individuals learn ways to reduce the physiological cues associated with anxiety and worry (Öst, 1987; Siev & Chambless, 2007)
  Interventions: Behavioral: Applied Relaxation (AR)
- Clinical monitoring control (Placebo Comparator): participants assigned to the clinical monitoring (CM) condition will receive the same information about the nature of GAD provided to participants in the active conditions ; however, they will not be randomized to treatment until after the 3-month follow-up assessment. To control for the effects of psychoeducation, symptom monitoring, contact by project staff, and maturation effects, participants will be asked to complete pre-, mid- and post-assessments, and will be informed that they will receive treatment.
  Interventions: Behavioral: Clinical Monitoring (CM)
- Combining the AMP and AR (Experimental): Both AMP and AR
  Interventions: Behavioral: Combining the AMP and AR

INTERVENTIONS:
Behavioral: AMP — The AMP is a computer-delivered attention modification protocol designed to enhance attention disengagement from threatening stimuli. The AMP protocol includes twelve 20-min sessions delivered over a 6-week period. During each session, participants will see 240 trials consisting of the various combinations of probe type (E or F), probe position (top or bottom), and word type (Neutral or Threat). 192 trials include one neutral word and one threat word: 2 (probe type) X 2 (probe position) X 2 (repetitions) X 24 (word pairs). On trials where participants see one neutral word and one threat word (i.e., 80% of the trials), the probe always follows the neutral word.
  Arms: 1 Attention Modification Program (AMP)
Behavioral: Applied Relaxation (AR) — Applied Relaxation (AR) is a behavioral, skills-based intervention where individuals learn ways to reduce the physiological cues associated with anxiety and worry (Öst, 1987; Siev & Chambless, 2007)
  Arms: Applied Relaxation (AR)
Behavioral: Clinical Monitoring (CM) — participants assigned to the clinical monitoring (CM) condition will receive the same information about the nature of GAD provided to participants in the active conditions
  Arms: Clinical monitoring control
Behavioral: Combining the AMP and AR — The AMP is a computer-delivered attention modification protocol designed to enhance attention disengagement from threatening stimuli. The AMP protocol includes twelve 20-min sessions delivered over a 6-week period. During each session, participants will see 240 trials consisting of the various combinations of probe type (E or F), probe position (top or bottom), and word type (Neutral or Threat). 192 trials include one neutral word and one threat word: 2 (probe type) X 2 (probe position) X 2 (repetitions) X 24 (word pairs). On trials where participants see one neutral word and one threat word (i.e., 80% of the trials), the probe always follows the neutral word. Applied Relaxation (AR) is a behavioral, skills-based intervention where individuals learn ways
  Arms: Combining the AMP and AR

SUMMARY:
Generalized Anxiety Disorder (GAD) has high prelevance (up to 8.5%; Roy-Byrne & Wagner, 2004) and leads to functional impairment (Wittchen et al., 2002; Ballenger et al., 2001). Researchers have demonstrated a relationship between attention bias to threatening information and GAD. However, this knowledge has not yet been translated into effective treatments. The goal of this project is develop and test a new computerized treatment for Generalized Anxiety Disorder.

DETAILED DESCRIPTION:
Generalized Anxiety Disorder (GAD) is characterized by excessive, uncontrollable worry (Barlow, et al., 1986) leading to medical over-utilization, poor perceived health, low ratings of quality of life, and impairment at work resulting in a significant economic and public health impact (Wittchen et al., 2002; Ballenger et al., 2001). Lifetime prevalence of GAD is high (5.7%, Kessler, et al, 2005), with even higher estimates in the primary care setting (8.5%, Roy-Byrne & Wager, 2004). Researchers have established a relationship between GAD and attention bias to threatening information (Mogg & Bradley 2005). This knowledge, however, has not been translated into more effective treatments for this disorder. This five-year, two site proposal aims to test a computerized treatment for GAD in a double-blind, placebo-controlled study bridging basic attention bias research and treatment outcome. We present the results from 7 studies demonstrating the efficacy of attention modification programs (AMP) in ameliorating symptoms of anxiety. Specifically, we report results from a pilot study of individuals with Generalized Anxiety Disorder (n=24, Dr Amir's lab), and high worries (n=24, Dr. Schmidt's lab) demonstrating the effectiveness of the procedures described in this proposal.

In brief, our intervention was effective in: a) changing biased attention, b) reducing symptoms of GAD, and c) maintaining its effects in up to one year follow-up. This technique for changing attention bias in GAD can provide a cost-effective and easy to administer treatment grounded in basic cognitive science that may help reduce suffering in individuals with anxiety. A larger study would allow us to test the treatment and examine the generalizability of the intervention to patients with GAD along with comorbid conditions. Moreover, we will examine the transportability of the intervention by examining the proposed intervention at two sites. There are currently 10 participants enrolled in the newest phase of pilot data collection (SDSU 6, FSU 4).

The goal of the current proposal is to extend these findings to a larger group of individuals with GAD and to examine the generalizability of the results to individuals with comorbid GAD. In the current proposal we will test two hypotheses:

1. Individuals with GAD completing the AMP will show a larger reduction in their attention bias to threat compared to the clinical monitoring group
2. Individuals with GAD completing AMP will show a larger reduction in anxiety symptoms compared to the clinical monitoring group.
3. Individuals with GAD completing AR will show a larger reduction in anxiety symptoms compared to the clinical monitoring group.

Specifically, in the current proposal directly responds to the NIMH priorities for evaluating user-friendly interventions and non-traditional delivery methods to increase access to evidence-based interventions. We will evaluate the efficacy of a 12-week computer-delivered home-based treatment program for GAD. Treatment will comprise a combination of two interventions shown to be efficacious in the treatment of GAD. The Attention Modification Program (AMP) is a computerized program designed to facilitate attention disengagement from threatening stimuli (Amir et al., 2009). Applied Relaxation (AR) is a behavioral, skills-based intervention where individuals learn ways to reduce the physiological cues associated with anxiety and worry (Öst, 1987; Siev & Chambless, 2007). Following the recommended guidelines of the NIMH Workgroup on Psychosocial Intervention Development (Hollon et al., 2002), we review evidence suggesting that both treatments are ideal candidates for the efficient, economical, and widespread transportation of evidence-based treatments for GAD. This proposal has the potential for a significant public health impact by evaluating a new method for delivering evidence-based interventions for hard-to-reach populations through the use of innovative technologies.

ELIGIBILITY:
Inclusion Criteria:

* Primary diagnosis of Generalized Anxiety Disorder

Exclusion Criteria:

* Evidence of suicidal intent
* Evidence of current substance abuse
* Evidence of current or past schizophrenia, bipolar disorder, or organic mental disorder
* Current CBT
* Change in other psychosocial or pharmacological treatment during the 12 weeks prior to study entry.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 193 (Actual)
Dates: Start 2007-12; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Hamilton Anxiety Rating Scale | Pre, Post, Followup

SECONDARY OUTCOMES:
Worry Domains Questionnaire | Pre, Post, Followup

CONTACTS AND LOCATIONS:
Overall Officials: Nader Amir, Ph.D., Principal Investigator — San Diego State University
Locations (1):
- San Diego State University, San Diego, California, United States

REFERENCES:
- [Derived] Amir N, Taboas W, Montero M. Feasibility and dissemination of a computerized home-based treatment for Generalized Anxiety Disorder: A randomized clinical trial. Behav Res Ther. 2019 Sep;120:103446. doi: 10.1016/j.brat.2019.103446. Epub 2019 Jul 26. PMID 31376708